CLINICAL TRIAL: NCT07374731
Title: Identification of Biomarkers of Risk for Pre-neoplastic and Neoplastic Lesions for the Development of Gastric Cancer
Acronym: DSCb score
Status: Recruiting | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2024-04
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigator propose the implementation of circulating biomarker monitoring, focusing on molecules related to the progression of gastric atrophy and/or associated with gastric cancer.

Monitoring these biomarkers will provide gastroenterologists with timely information on individuals at risk and, if values worsen during follow-up, will alert physicians observing these patients to evaluate them.

This monitoring will be offered to individuals who contact the IBO (Immunopatologia e Biomarcatori Oncologici) Unit at CRO (Centro di Riferimento Oncologico) in Aviano requesting an assessment of gastric function through pepsinogen and G17 gastrin level testing. Monitoring these biomarkers will provide a dynamic analysis of patients' gastric status, allowing for timely intervention in case of deviations from normal values. This proactive approach is important for the preventive management of gastric diseases, particularly for the diagnosis and monitoring of gastric atrophy and gastric cancer.

The IBO unit of the CRO in Aviano, together with the pathological anatomy and clinical units of gastroenterology, medical oncology, and surgery, will play a role in coordinating and implementing this monitoring program, thus contributing to the promotion of gastric health and the prevention of associated diseases.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18;
* Ability to understand, accept, and sign the informed consent form for the study;
* Ability to understand, accept, and sign the consent form for data processing;
* Ability to understand, accept, and sign the consent form for the collection of a serum sample for research purposes;
* Patients who are fasting and have requested a pepsinogen test or gastroscopy, or who have gastric cancer prior to treatment;
* Subjects who are fasting and have suspected pre-neoplastic/neoplastic gastric lesions or who have requested a pepsinogen test and for whom endoscopic examination data are available.

Exclusion Criteria:

* Patients under the age of 18
* Pregnant women
* Patients with a coexisting or previous diagnosis of another malignant neoplasm in the last 5 years
* Patients unable to understand, accept, and sign the consent form for data processing

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be divided into two patient cohorts:
  * a retrospective cohort comprising biological material (serum) stored at the IBO unit of the CRO in Aviano and/or at the Biobank since 2014 from subjects with suspected gastric lesions or gastric cancer;
  * a prospective cohort of subjects with prescriptions for pepsinogen and G17 gastrin testing. Selection will be made from among those who present at the CRO blood collection room in Aviano, in gastroenterology, or who are admitted to medical oncology or surgery for gastric cancer. Hospitalized patients will undergo fasting blood sampling before therapy or surgery. Subjects belonging to high-risk categories or diagnosed with neoplasia will undergo a second blood sampling during follow-up to monitor any disease progression or therapeutic response.
Sampling Method: Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2025-05-21 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the association between the levels of selected biomarkers and the diagnosis obtained after endoscopic examination and histological evaluation of the biopsies taken. | 36 months
  The mean value of biomarkers level in positive and negative biopsy will be evaluated

SECONDARY OUTCOMES:
Evaluate the prognostic potential of baseline levels of the biomarkers analyzed | 36 months
  Mean difference of biomarkers between responders and non responders
Identify biomarkers with the best relation with more advanced pre-neoplastic conditions and with neoplasia. | 36 months
  Mean difference of biomarkers level in subgroups of patients with the condition under investigation
Compare the predictive accuracy of risk between the DSCb test and the DSCb test with the addition of the best-performing biomarker | 36 months
  Accuracy will be calculated as number of patients correctly classified over the total number of patients.
Monitor test values during follow-up in subjects classified as high risk to assess the possible progression of the pre-neoplastic lesion | 36 months
  Likelihood ratio of the two tests will be reported
Monitor test values during follow-up in subjects with neoplasia to assess the potential of the test in therapeutic response | 36 months
  Test will be compared by mean of ROC curve analysis

CONTACTS AND LOCATIONS:
Overall Officials: Valli De Re, Principal Investigator — Centro di Riferimento Oncologico
Locations (1):
- Centro di Riferimento Oncologico (CRO) di aviano-IRCCS, Aviano, Pordenone, Italy